CLINICAL TRIAL: NCT07303881
Title: A Clinical Study Evaluating the Safety and Efficacy of Golidocitinib in Patients With Refractory Immune-related Hematologic Toxicities of Advanced Lung Cancer
Brief Title: Golidocitinib for Refractory Immune-related Hematologic Toxicities of Advanced Lung Cancer
Acronym: JACKPOT22
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Director, Head of Thoracic Surgery, Principal Investigator, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-244-02
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: IrAE; Hematologic Disorder; Lung Cancer (Locally Advanced or Metastatic)
Keywords: Immune-related hematologic toxicities; irAE; Lung cancer
MeSH Terms: conditions — Hematologic Diseases; Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golidocitinib (Experimental): Based on the BOIN dose escalation and Simon two-stage efficacy assessment design, if the dose of golidocitinib used in Part B is 75 mg, the total number of subjects to be included in Parts A and B is 10; if the dose of golidocitinib used in Part B is 150 mg, the total number of subjects to be included in Parts A and B is 13-16.
  Interventions: Drug: golidocitinib

INTERVENTIONS:
Drug: golidocitinib — Golidocitinib treatment can be discontinued once clinical remission is achieved, with a maximum maintenance period of 12 weeks.

SUMMARY:
This study is a single-arm clinical trial designed to evaluate the safety and efficacy of golidocitinib in patients with refractory, immune-related hematologic toxicity in advanced lung cancer.

DETAILED DESCRIPTION:
This is a single-center, single-arm clinical trial designed to evaluate the safety and efficacy of golixitinib in patients with advanced lung cancer exhibiting refractory immune-related hematologic toxicity. In this study, refractory immune-related hematologic toxicity was defined as grade ≥3 hematologic toxicity in patients with advanced lung cancer receiving immune checkpoint inhibitor therapy, unresponsive to treatment with hormones/hematopoietic factors/blood transfusions, and with a positive antinuclear antibody (ANA) profile (anti-SSA antibody). Patients with refractory immune-related hematologic toxicity will primarily receive golixitinib. This study comprises two parts:

Part A (dose escalation): This part will include patients with refractory immune-related hematologic toxicity to determine the safety and initial hematologic toxicity mitigation of golixitinib in this population, and to determine the recommended dose for Part B (dose extension).

Part B (dose extension): This part will include patients with refractory immune-related hematologic toxicity to further explore the hematologic toxicity mitigation and safety of the selected dose of golixitinib in this population.

Based on the BOIN dose escalation and Simon two-stage efficacy assessment design, if the dose of golixitinib used in Part B is 75 mg, the total number of subjects to be included in Parts A and B is 10; if the dose of golixitinib used in Part B is 150 mg, the total number of subjects to be included in Parts A and B is 13-16.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated informed consent form, including compliance with the Informed Consent Form (ICF) and the requirements and limitations listed in this protocol.
2. The subject is ≥18 years of age at the time of signing the ICF.
3. Has not experienced disease progression in the past two weeks and has a Eastern Cooperative Oncology Group (ECOG) score of 0-2, with a predicted survival of ≥12 weeks.
4. Pathologically or cytologically confirmed locally advanced (American Joint Committee on Cancer, AJCC 8th edition IIIB and IIIC stages) or metastatic (stage IV) non-small cell lung cancer, or extensive-stage small cell lung cancer (AJCC 8th edition TNM staging of lung cancer stage IV, or T3-4 disease caused by multiple pulmonary nodules with excessive disease spread, or tumor/nodule size too large for a tolerable radiation therapy plan).
5. Patients confirmed by an accredited local laboratory to lack any therapeutically targeted driver gene mutations, i.e., driver gene-negative subjects.
6. Patients experiencing grade ≥3 refractory hematologic toxicity (white blood cell count <2.0 × 10⁹/L or/and absolute neutrophil count <1.0 × 10⁹/L or/and platelet count <50 × 10⁹/L or/and hemoglobin <8.0 g/dL, specific hematologic parameters are detailed in Appendix D), during treatment with immune checkpoint inhibitors (including monotherapy or combination therapy), and the toxicity is considered to be immune-related. Refractory toxicity is defined in two main ways: ① Resistance to conventional treatment: No significant improvement in hematologic toxicity after at least 3 days of supportive care including the use of hormones (e.g., methylprednisolone ≥1 mg/kg/d), hematopoietic growth factors (e.g., G-CSF, TPO), and/or blood transfusions; ② Positive antinuclear antibody profile indicating anti-SSA antibodies and/or Ro52 antibodies, suggesting an immune-mediated mechanism.
7. Patients with brain metastases must be asymptomatic or have been treated and have stable disease after discontinuation of steroids and anticonvulsants. Patients suspected of having brain metastases at screening should undergo brain CT/MRI before study enrollment.
8. At least one measurable lesion (as defined in RECIST 1.1): a lesion that has not undergone radiotherapy, has a long diameter ≥10 mm (short diameter ≥15 mm for lymph node lesions), and can be accurately and repeatedly measured from baseline on CT or MRI; and a measurable lesion outside the central nervous system.
9. Adequate organ system functional reserve, summarized as follows:

   * Total bilirubin ≤1.5×ULN; if Gilbert's syndrome (unconjugated hyperbilirubinemia) is present, total bilirubin should be ≤3×ULN.
   * ALT and AST ≤2.5×ULN. For patients with documented liver metastases, AST and ALT levels ≤5×ULN.
   * Creatinine clearance, calculated using the Cockcroft-Gault method, >60 ml/min for patients treated with cisplatin and >45 ml/min for patients treated with carboplatin.
   * Urinalysis shows less than 2+ protein in urine, or 24-hour urine protein quantification <1g.
   * Good coagulation function, defined as International Normalized Ratio (INR) and/or Prothrombin Time (PT) ≤1.5 times the ULN and/or Activated Partial Thromboplastin Time (APTT) ≤1.5 of the upper limit of normal; if the subject is receiving anticoagulation therapy, PT is acceptable as long as it is within the range intended for use with the anticoagulant.
   * Serum amylase ≤1.5 times the ULN and/or serum lipase ≤1.5 times the ULN.
   * Echocardiography (ECHO) shows a left ventricular ejection fraction (LVEF) ≥55%.
10. Women of Childbearing Potential (WOCBP) must undergo a urine and/or serum pregnancy test (if the urine test cannot confirm a negative result) within 7 days prior to the first dose of the study drug, and the result must be negative; WOCBP or male subjects and their WOCBP partners should agree to use effective contraception from the signing of the ICF until 6 months after the last dose of the study drug. k. Participants should be able to understand the study protocol and voluntarily comply with the study and follow-up.

Exclusion Criteria:

a. An active autoimmune disease requiring systemic treatment (e.g., use of disease-modifying medications, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatment.

b. Prior to the first dose, any other form of immunosuppressive therapy other than corticosteroids (e.g., TNF-α inhibitors, mycophenolate mofetil, gamma globulin, rituximab, other JAK inhibitors, etc.) was received for hematologic toxicity.

c. Spinal cord compression or meningeal metastases are present. d. Any of the following medical histories:

* Currently participating in an interventional clinical trial, or having received other investigational drugs or used investigational devices within 4 weeks prior to the first dose; any drug still in development requires a 5-half-life washout (or discussion with the research team);
* Underwent major surgery (excluding diagnostic or biopsy, excluding vascular access) within 4 weeks prior to the first dose, or is expected to undergo major surgery during the study;
* Received palliative radiation therapy within 2 weeks prior to the first dose;
* Have experienced a serious arterial/venous thrombotic event within 6 months prior to the first dose, including cerebrovascular accidents (e.g., history of stroke or intracranial hemorrhage), deep vein thrombosis, and pulmonary embolism;
* Currently receiving (or unable to discontinue at least 1 week prior to the first dose) any known potent inducer or inhibitor of CYP3A, herbal supplements, or foods;
* Have experienced a grade CTCAE > 1 adverse event (excluding any degree of alopecia and hematologic toxicity) due to prior treatment prior to the first dose. e. Has received a solid organ or blood system transplant (e.g., a previous allogeneic bone marrow transplant).

  f. Has a history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring corticosteroid therapy, or currently has active interstitial lung disease (including interstitial lung changes), or immune-mediated pneumonitis caused by immunotherapy.

  g. Has been diagnosed with another malignancy within 5 years prior to the first dose, excluding clinically cured basal cell carcinoma, squamous cell carcinoma, and/or radically resected carcinoma in situ.

  h. Has received a live vaccine, including attenuated live vaccines, excluding inactivated vaccines, within 30 days prior to the first dose.

  i. Has known active tuberculosis, such as a positive tuberculin (PPD) test (induration diameter > 10 mm), a positive T-SPOT test, tuberculous lesions on chest X-ray/CT, or other positive results found according to routine clinical screening (excluding those cured by investigator assessment after standard anti-tuberculosis treatment).

  j. Subjects with pre-existing, uncontrollable severe infectious diseases must be excluded. If an infectious disease occurred within two months prior to the first dose, its control must be assessed by the research team to determine eligibility for enrollment.

  k. Subjects with active infections, including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) (see table below), and active COVID-19 infection (determined by the investigator to be clinically significant, with signs or symptoms). COVID-19 testing will be based on local practice.

  l. Meeting any of the following cardiac criteria:
* Congestive heart failure (CHF) classified as >II by the New York Heart Association (NYHA);
* Clinically significant valvular heart disease, hypertrophic or constrictive cardiomyopathy;
* Any clinically significant abnormality on resting ECG, such as complete left bundle branch block, second/third-degree atrioventricular block, or PR interval >250 msec;
* Average calibrated QTcF >470 msec on three resting ECGs during the screening period;
* Any factor that could increase the risk of QT interval prolongation or arrhythmic events (e.g., heart failure, hypokalemia, congenital long QT syndrome, or a first-degree relative with long QT syndrome or a family history of unexplained sudden death under 40 years of age, or any concomitant medication known to prolong the QT interval);
* Ventricular arrhythmias requiring treatment;
* An acute myocardial infarction (AMI), the onset of unstable angina, or a new onset of angina within 6 months prior to administration.

  m. Hypersensitivity to the study drug or any component thereof. n. Intractable nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing medication, intestinal obstruction, or a history of bowel resection that may prevent adequate absorption of the study drug.

  o. Pregnancy or lactation. p. Known bleeding diathesis, i.e., hemophilia or von Willebrand disease. q. Investigator assessment indicating a serious or uncontrolled systemic disease (including poorly controlled hypertension and bleeding disorders) that precludes participation in the clinical study or may lead to poor adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate of immune-related hematologic toxicities | 12 weeks
  The proportion of subjects who achieved clinical remission of immune-related hematologic toxicities treated with golidocitinib (clinical remission is defined as a degraded hematologic toxicity grade within 1 week of golidocitinib use, a hematologic toxicity grade ≤1 within 2 weeks, and no relapse before discontinuation of treatment). This was assessed by the investigator based on laboratory indicators and the subject's clinical condition.

SECONDARY OUTCOMES:
Negative conversion rate of SSA/Ro52 antibody | 12 weeks
  The proportion of subjects whose SSA/Ro52 antibody test results changed from positive to negative. This was assessed by the investigator based on laboratory indicators and the subjects' clinical condition.
Progression free survival | 2 years
  The duration from the start of immunotherapy to disease progression or death from any cause as determined by RECIST 1.1, regardless of whether the subject discontinued the investigational drug or received other anticancer treatments before disease progression. This assessment is conducted by the investigator based on the subject's imaging and clinical condition.
Overall survival | 2 years
  The time from the start of immunotherapy to the subject's death from any cause, regardless of whether the subject received other anticancer treatments. Assessed by the investigator based on the subject's clinical condition.
Adverse events | 12 weeks
  Incidence of adverse events/serious adverse events, severity as assessed by CTCAE v5.0, and relevance to the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data will be kept confidential before publication.